CLINICAL TRIAL: NCT00758004
Title: An Open Label, Randomized, Single Dose, Two-Way Crossover Bioequivalence Study Comparing A New 80 Mg (2x40 mg) Pediatric Appropriate Formulation To A 80 Mg Commercial Atorvastatin Calcium Tablet Formulation In Healthy Subjects
Brief Title: Bioequivalence Study Of Pediatric Appropriate Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A2581175
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia
Keywords: Cardiovascular Diseases
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (Other): Commercial 80 mg atorvastatin tablet
  Interventions: Drug: Atorvastatin
- Test (Other): Pediatric appropriate atorvastatin 40mg formulation
  Interventions: Drug: Atorvastatin pediatric appropriate formulation

INTERVENTIONS:
Drug: Atorvastatin — A single dose of 80 mg atrovastatin tablet
  Arms: Reference
Drug: Atorvastatin pediatric appropriate formulation — A single dose of pediatric appropriate atorvastatin 80 mg formulation
  Other Names: Atorvastatin
  Arms: Test

SUMMARY:
To determine bioequivalence of pediatric appropriate 80 mg atorvastatin formulation comparing to the 80 mg commercial atorvastatin calcium tablet formulation.

DETAILED DESCRIPTION:
Determination of Bioequivalence

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female volunteers
* Mass Index (BMI) of approximately 18 to 30 kg/m2

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* A positive urine drug screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Primary study endpoints will be AUClast, AUCinf (if data permit) and Cmax from plasma atorvastatin concentration data. | 5 months

SECONDARY OUTCOMES:
Secondary endpoints will include Tmax and t1/2 (if data permit) of atorvastatin ; AUClast, AUCinf, Cmax, Tmax, and t1/2 (if data permit) of o-hydroxyatorvastatin and p-hydroxyatorvastatin. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581175&StudyName=Bioequivalence%20Study%20Of%20Pediatric%20Appropriate%20Formulation